CLINICAL TRIAL: NCT06882993
Title: Feasibility of a Minimally Invasive Diagnostic Algorithm in Suspected Crohn's Disease - a Prospective Comparison of Pan-Enteric Capsule Endoscopy Versus Ileocolonoscopy Plus MR Enterography or Small-Bowel Capsule Endoscopy
Brief Title: Feasibility of a Minimally Invasive Diagnostic Algorithm in Suspected Crohn's Disease
Acronym: ANDI-3
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Esbjerg Hospital - University Hospital of Southern Denmark (Other)
Collaborators: Odense University Hospital (Other); Svendborg Hospital (Other); Skane University Hospital (Other); Vejle Hospital (Other)
Responsible Party: Principal Investigator, Frederik Drejer Thrane, PhD Student, Esbjerg Hospital - University Hospital of Southern Denmark
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 24/50881
Record Dates: First submitted 2025-02-26; First posted 2025-03-19 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Crohn's Disease
Keywords: capsule endoscopy; panenteric capsule endoscopy; Crohn's disease; inflammatory bowel disease
MeSH Terms: conditions — Crohn Disease; Inflammatory Bowel Diseases | interventions — Endoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Minimally invasive diagnostic algorithm (Experimental)
  Interventions: Diagnostic Test: Panenteric capsule endoscopy
- Traditional work-up (Active Comparator): Colonoscopy and either MRI enterography or small bowel capsule endoscopy
  Interventions: Diagnostic Test: Ileocolonoscopy; Diagnostic Test: MRI enterography; Diagnostic Test: Small bowel capsule endoscopy

INTERVENTIONS:
Diagnostic Test: Panenteric capsule endoscopy — Panenteric capsule endoscopy
  Arms: Minimally invasive diagnostic algorithm
Diagnostic Test: Ileocolonoscopy — Endoscopic examination of the colon and terminal ileum after bowel preparation.
  Arms: Traditional work-up
Diagnostic Test: MRI enterography — MRI of the small bowel
  Arms: Traditional work-up
Diagnostic Test: Small bowel capsule endoscopy — Capsule endoscopy of the small bowel
  Arms: Traditional work-up

SUMMARY:
The goal of this clinical trial is to learn whether a camera pill examination of the whole bowel can be used to diagnose Crohn's disease instead of colonoscopy and a small bowel examination (either MRI or camera pill) in patients aged 18-40 years suspected of having Crohn's disease.

The main question it aims to answer is:

How many patients examined with a camera pill examination of the whole bowel will have a complete examination of the whole bowel and have a diagnosis made without need for any more examinations?

Researchers will compare with patients examined with colonoscopy and a small bowel examination.

Participants will:

* Be examined with either a camera pill examination of the whole bowel, or a colonoscopy and a small bowel examination
* Have their electronic medical records checked to see if a diagnosis has been made
* Have an interview every three months if diagnosed with an inflammatory bowel disease or after a year if no disease was found

ELIGIBILITY:
Inclusion Criteria:

* Clinical suspicion of CD*
* Age 18-40 years
* Signed informed consent

  *A clinical suspicion of CD is based on the following definition:
* Diarrhea and/or abdominal pain for more than 1 month (or repeated episodes of diarrhea and/or abdominal pain) and either

  * fecal calprotectin ≥ 200 mg/kg or
  * fecal calprotectin ≥ 50 mg/kg plus one or more of the following findings:
* C-reactive protein (CRP) > 5 mg/L
* Thrombocytosis (> 400 x 109/L)
* Anemia (hemoglobin < 7.0 mmol/L for women and < 8.0 mmol/L for men or a decrease > 0.5 mmol/L compared to the usual level)
* Prolonged fever (> 37.5 ◦C for more than 2 weeks)
* Weight loss (≥ 3 kg or ≥ 5% compared to the normal body weight)
* Perianal abscess / fistula
* Family history of inflammatory bowel disease.

Exclusion Criteria:

* Previous intestinal resection
* Positive serologic markers for celiac disease
* Positive stool polymerase chain reaction for pathogenic bacteria
* Positive stool polymerase chain reaction for intestinal parasites
* Suspected or established acute bowel obstruction (ileus)
* Intake of NSAIDs or acetylsalicylic acid ≤ 4 weeks before inclusion, except low-dose, prophylactic acetylsalicylic acid (≤ 150 mg per day)
* Intake of opioid or opioid-like medications ≤ 1 week before inclusion
* Pregnancy or lactation
* Inability to comply with protocol requirements, e.g. for reasons including alcohol or recreational drug abuse
* Known gastrointestinal disorder other than functional gastrointestinal disorders
* Renal failure defined by a plasma-creatinine above the normal reference range

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 165 (Estimated)
Dates: Start 2025-02-26 (Actual); Primary Completion 2027-08-31 (Estimated); Study Completion 2028-08-31 (Estimated)

PRIMARY OUTCOMES:
Diagnostic completeness | Immediately after initial diagnostic procedure
  Proportion of patients in each arm achieving a complete gastrointestinal assessment and an unambiguous diagnosis after completion of the initial diagnostic procedure(s) without need for supplementary examinations

SECONDARY OUTCOMES:
Feasibility of pan-enteric CE | After completion of follow-up (12 months)
  Number of patients with suspected CD examined with pan-enteric CE and the number of ICs avoided
Additional examinations | After completion of follow-up (12 months)
  Need for additional examinations in the two randomization arms
Safety | After completion of follow-up (12 months)
  Number of severe adverse events
Time to diagnosis | After completion of follow-up (12 months)
  Time from referral or first diagnostic procedure to final diagnosis and treatment
Disease classification and medical treatments | After completion of follow-up (12 months)
  Disease classification and medical treatments in the two randomization arms
Patient satisfaction | Immediately after initial diagnostic procedure
  Difference in Gastrointestinal Endoscopy Satisfaction Questionnaire (GESQ) score
Costs | After completion of follow-up (12 months)
  Expenditure on diagnostic procedures, treatment and loss of productivity
Artificial intelligence | Immediately after initial diagnostic procedure
  Diagnostic utility of AI algorithms in detection of gastrointestinal pathology using pan-enteric CE - sensitivity, specificity, severity, prediction and impact on clinical decision making

CONTACTS AND LOCATIONS:
Overall Officials: Frederik D Thrane, MD, Principal Investigator — Esbjerg Hospital - University Hospital of Southern Denmark
Locations (5):
- Denmark (4):
  - Esbjerg Hospital - University Hospital of Southern Denmark, Esbjerg
  - Odense University Hospital, Odense C
  - Odense University Hospital - Svendborg Hospital, Svendborg
  - Lillebaelt Hospital Vejle - University Hospital of Southern Denmark, Vejle
- Skåne University Hospital, Malmo, Sweden

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR

DOCUMENTS (1):
  • Study Protocol (2024-11-08): https://cdn.clinicaltrials.gov/large-docs/93/NCT06882993/Prot_000.pdf